CLINICAL TRIAL: NCT07104929
Title: Prospective Human Study Evaluating the Effects of Beta Glucan 500 on Markers of Biological Age and Immune Age: An Open-label Pilot Study
Brief Title: Beta Glucan 500 and Biological Age and Immune Age
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OvationLab (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BWH-002
Record Dates: First submitted 2025-07-28; First posted 2025-08-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Aging
Keywords: aging; biological age; immunosenescence; beta glucan
MeSH Terms: interventions — beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beta Glucan (Experimental)
  Interventions: Dietary Supplement: Beta Glucan

INTERVENTIONS:
Dietary Supplement: Beta Glucan — 12 weeks of supplementation with two capsules daily of BWH Labs Beta Glucan 500

SUMMARY:
The primary purpose of this study is to evaluate the effects of BWH Labs - Beta Glucan 500 on biomarkers of biological and immune age among healthy adults.

A single-arm, open-label prospective study will be conducted evaluating the impact of 12 weeks of supplementation with two capsules daily of Beta Glucan 500 on a variety of validated markers of biological and immune age on the comprehensive TruAge panel (TruDiagnostics, Lexington, KY).

ELIGIBILITY:
Inclusion Criteria:

1. Adult females or males age ≥ 40 years
2. Ability to read and speak English
3. Previous completion of a TruDiagnostic TruAge test within the past three months to enable comparison of previous biomarkers to the same biomarkers after intervention
4. DunedinPACE estimate of aging >0.9

Exclusion Criteria:

1. Current diagnosis and treatment for an autoimmune condition
2. Current use of beta-glucan or mushroom dietary supplement
3. Known allergies to beta glucan, yeast, or mushrooms
4. Currently pregnant or lactating women or women planning to become pregnant in the next 12 weeks
5. Current diagnosis of a chronic health condition (e.g., cancer, heart failure, history of pancreatitis, type I or II diabetics on insulin) deemed clinically contraindicated for the study protocol
6. Participants unable to provide consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Testing | Change from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- OvationLab, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Private genetic and epigenetic data